CLINICAL TRIAL: NCT07012200
Title: Exploring the Effect of Immersive Interactive Nursing Guidance on Anxiety, Cognition and Self-efficacy in Patients With Coronary Heart Disease Undergoing Cardiac Catheterization
Brief Title: Effect of Immersive Interactive Nursing Guidance on Anxiety, Cognition, and Self-efficacy in CHD Patients Undergoing Cardiac Catheterization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to reduced bed capacity in the cardiology ward, insufficient nursing manpower, hospital accreditation preparation, and exhaustion of platform budget. 112 participants were recruited; final analysis included 108.
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 111-208-E
Record Dates: First submitted 2023-08-27; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-03

CONDITIONS: Augmented Reality; Nursing Education; Anxiety; Immersive
Keywords: cardiac catheterization; immersive Interactive; Nursing Guidance
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immersive Interactive Nursing Instruction (Experimental): Immersive interactive nursing guidance, which includes: 360-degree introduction to the environment of the cardiac catheterization laboratory, cardiac catheterization procedures (including preoperative, intraoperative, and postoperative), wound care, and precautions for home care (including diet, medication, and exercise)
  Interventions: Other: Immersive Interactive Nursing Instruction
- Routine Nursing Instructions (Active Comparator): Health education by talking and leaflets and key explanations, and providing talks and consultations
  Interventions: Other: Routine Nursing Instructions

INTERVENTIONS:
Other: Immersive Interactive Nursing Instruction — 360-degree introduction to the environment of the cardiac catheterization laboratory, cardiac catheterization procedures (including preoperative, intraoperative, and postoperative), wound care, and precautions for home care (including diet, medication, and exercise)
  Arms: Immersive Interactive Nursing Instruction
Other: Routine Nursing Instructions — Health education by talking and leaflets and key explanations, and providing talks and consultations
  Arms: Routine Nursing Instructions

SUMMARY:
The purpose of this study is to explore the effect of immersive interactive nursing guidance on anxiety, disease cognition, self-efficacy and satisfaction in patients undergoing cardiac catheterization for coronary heart disease. It will help clinical medical staff understand the timing and effectiveness of interventional immersive interactive nursing guidance for patients undergoing cardiac catheterization. Therefore, the research hypotheses to be verified in this study are as follows:

1. There are differences in anxiety between patients receiving immersive interactive nursing guidance and traditional written medical education for cardiac catheterization.
2. There are differences in disease cognition between patients receiving immersive interactive nursing guidance and traditional written health education for cardiac catheterization.
3. There are differences in the self-efficacy of patients receiving immersive interactive nursing guidance and traditional written medical education for cardiac catheterization.
4. There are differences in the satisfaction with the use of immersive interactive nursing guidance.

DETAILED DESCRIPTION:
The subjects of this study are patients who received cardiac catheterization for the first time. The experimental study was conducted with a single-blind study design. The experimental group used immersive interactive nursing guidance and the control group used general nursing guidance to conduct a comparative study of different nursing guidance before discharge. . The researcher first makes a random admission form. For those who meet the research admission conditions, the researcher first gives an explanation, obtains the patient's consent and signs the consent form for the human experiment, and assigns the research cases to the experimental group and the control group according to random acceptance. A structured questionnaire was used to investigate the differences in the degree of improvement in anxiety, cognition and self-efficacy of patients with coronary heart disease before they were discharged from the hospital after cardiac catheterization. After filling in the basic information on the day of admission, the patient began to fill in the pre-test questionnaires: "Situation and Trait Anxiety Scale", "Cognition Scale", and "Self-Efficacy Scale". After the pre-test questionnaires were collected, the experimental group received immersive interactive nursing guidance in addition to general routine nursing guidance (general routine nursing health education leaflets, combined with oral health education and key explanations, talks and consultations), which included : 360-degree introduction to the environment of the cardiac catheterization laboratory, cardiac catheterization process (including preoperative, intraoperative, and postoperative), wound care, precautions for home care (including diet, medicine, and exercise), and nursing guidance content about 12-15 minutes long , can be watched by mobile phone or tablet, and can be watched repeatedly and experience interactive nursing guidance according to the patient's needs. The two groups of patients completed the "Situation and Trait Anxiety Scale (Post-test)" after nursing guidance and before performing cardiac catheterization; it did not affect the patient's rest, stable condition and completion of the "Cognitive Scale (Post-test)" and "Self-Test Scale" before discharge. Efficacy Scale (Post-test)" and Satisfaction Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 years or older with clear consciousness
* Diagnosed with coronary artery disease by a cardiologist and undergoing first-time cardiac catheterization or treatment
* Able to communicate in Mandarin or Taiwanese, and literate

Exclusion Criteria:

* Diagnosed with unstable coronary artery disease or acute myocardial infarction
* Requiring emergency cardiac catheterization or treatment

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
anxiety index | within 24 hours after admission and prior to catheterization
  Situation and Trait Anxiety Inventory,Score range 20-80 points,Higher scores indicate higher levels of anxiety.
cognitions | within 24 hours after admission and prior to catheterization
  Self-made cardiac catheterization cognition questionnaire, the scale includes what is cardiac catheterization, complications, precautions for cardiac catheterization, drug use, social activities, daily care, etc. The higher the score, the higher the awareness
Self-efficacy | within 24 hours after admission and prior to catheterization
  General Self-Efficacy Scale,10 items, each item is scored with 1 point for completely incorrect, 2 points for somewhat correct, 3 points for most correct, 4 points for completely correct, the higher the score, the higher the self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No